CLINICAL TRIAL: NCT07178418
Title: The Effects of a Muscle Architecture-Based Exercise Program and the Alfredson Protocol on Muscle-Tendon Architecture and Physical Performance in Subjects With Achilles Tendinopathy
Brief Title: Muscle Architecture vs Alfredson Protocol in Achilles Tendinopathy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Halic University (Other)
Collaborators: Istanbul University (Other)
Responsible Party: Principal Investigator, Ömer Bayrak, Research Assistant, Halic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Muscle Architecture
Record Dates: First submitted 2025-09-02; First posted 2025-09-17 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Achilles Tendinopathy (AT); Eccentric Exercise Training; Muscle Architecture; Isokinetic Test; Ultrasound; Balance; Anaerobic Power
Keywords: Achilles tendinopathy; muscle architecture; isokinetic strength; Alfredson protocol; tendon architecture

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Alfredson protocol (Active Comparator): Participants in this group will follow the classical Alfredson eccentric heel-drop protocol, widely used in the management of Achilles tendinopathy.
  Interventions: Other: Alfredson Protocol
- muscle architecture-based exercise program (Experimental): Participants in this group will perform an exercise program tailored to the architectural properties of the triceps surae muscles. Positioning and loading strategies will be individualized to optimize activation of the soleus and gastrocnemii.
  Interventions: Other: Muscle Architecture-Based Exercise Program

INTERVENTIONS:
Other: Muscle Architecture-Based Exercise Program — Participants in this arm will perform exercises specifically designed according to the architectural and functional properties of the triceps surae muscles. For example, knee-flexed positions will be used to target the soleus, while knee-extended positions will be emphasized for the gastrocnemii. Loading intensity and exercise progression will be tailored to optimize tendon and muscle remodeling.
  Arms: muscle architecture-based exercise program
Other: Alfredson Protocol — This intervention involves the traditional eccentric heel-drop program, originally developed for mid-portion Achilles tendinopathy. Participants perform three sets of 15 repetitions, twice daily, throughout the intervention period. Exercises are carried out both with the knee extended and flexed to load different portions of the triceps surae. The protocol applies repetitive eccentric loading to the Achilles tendon with the aim of stimulating collagen synthesis, reducing symptoms, and promoting tendon adaptation.
  Arms: Alfredson protocol

SUMMARY:
Achilles tendinopathy is a frequent overuse disorder caused by repetitive loading of the tendon, particularly observed in athletes and middle-aged men. It is typically characterized by mid-portion pain, stiffness in the morning, and functional limitations, with structural alterations such as thickening and disrupted collagen alignment. Chronic progression often compromises performance and quality of life.

Eccentric training protocols, such as the Alfredson regimen, are commonly prescribed but their standardized nature does not fully address individual variability. Alternative approaches including Heavy Slow Resistance training and progressive loading models (e.g., Silbernagel protocol) have demonstrated clinical effectiveness and higher patient adherence, yet they still apply uniform loading across the triceps surae without accounting for architectural differences.

Given the heterogeneous structure of the soleus and gastrocnemii, targeted loading strategies may be required to optimize tendon adaptation. To address this, the present study employs a muscle architecture-based exercise program tailored to the functional and structural properties of each muscle. Ultrasound imaging will be used to evaluate muscle-tendon morphology, while isokinetic dynamometry and functional performance tests will quantify outcomes. Pain (VAS) and functional capacity (VISA-A) will also be assessed.

This randomized controlled trial aims to compare the effectiveness of an architecture-specific program with the Alfredson protocol on tendon remodeling, strength, endurance, functional performance, and symptom reduction in individuals with non-insertional Achilles tendinopathy.

DETAILED DESCRIPTION:
Achilles tendinopathy is an overuse injury that develops as a result of repetitive microtrauma and is commonly observed in athletes as well as in sedentary male individuals. The clinical presentation is typically characterized by localized pain in the mid-portion of the tendon, tenderness, morning stiffness, and symptoms exacerbated by activity. Structurally, the condition is associated with tendon thickening, reduced echogenicity, and disorganization of collagen alignment . As the pathology becomes chronic, a marked decline in functional capacity is observed, which negatively affects both athletic performance and quality of life.

Conservative management is recommended as the first line of treatment, with the eccentric exercise protocol being the most widely used approach. Developed by Alfredson et al. (1998), this protocol consists of performing three sets of fifteen repetitions twice daily, aiming to stimulate collagen synthesis by mechanically loading the tendon. However, studies have shown that this protocol is not effective in every case; in some individuals, symptoms persist, and because the loading scheme is standardized, it fails to account for inter-individual variability. As an alternative, the Heavy Slow Resistance (HSR) exercise protocol, which includes both eccentric and concentric contractions, is applied three times per week. By incorporating controlled, high-resistance, slow-tempo loading, it aims to achieve functional recovery. Studies by Beyer et al. (2015) demonstrated that the HSR protocol yields clinical outcomes comparable to those of the Alfredson protocol, with higher patient satisfaction and compliance. In addition, the protocol developed by Silbernagel et al. (2007) incorporates both eccentric and concentric loading as well as functional activities in a more progressive model. By tailoring exercises to symptom tolerance during the acute and subacute phases and integrating plyometric activities such as hopping and jumping in the later stages, this protocol adopts a function-oriented perspective. Other conservative interventions, including extracorporeal shock wave therapy, cryotherapy, transverse friction massage, and footwear modifications, may provide symptomatic relief; however, their contribution to tendon remodeling is limited, and they do not ensure long-term structural or functional recovery. Although the Alfredson, HSR, and Silbernagel protocols are clinically effective, they carry significant limitations as they are not designed with muscle architecture-specific loading strategies.

The triceps surae muscle group exhibits heterogeneity in terms of architecture and function: the soleus muscle, with relatively short fascicle length, large cross-sectional area, and high pennation angle, contributes primarily to stability and endurance; the medial gastrocnemius is involved in both stability and controlled force generation; and the lateral gastrocnemius, with long fascicles and a narrow pennation angle, plays a key role in explosive force production. Despite these structural differences, both HSR and Silbernagel protocols apply a uniform loading strategy across all triceps surae muscles. For instance, optimal activation of the soleus requires the knee to be flexed, whereas activation of the medial and lateral gastrocnemius requires knee extension. Some existing protocols fail to consider such joint positioning, which may result in deviations from the optimal contraction axis, thereby reducing the effectiveness of muscle activation. This limitation may create uncertainty in the distribution of loading stimuli, hindering adequate tissue adaptation.

The muscle architecture-based exercise program to be implemented in this study is specifically designed in accordance with the architectural characteristics of each muscle, with the aim of providing the most optimal stimulus for each. Muscle and tendon architecture will be assessed using ultrasonography; strength outcomes will be measured with an isokinetic dynamometer; and functional performance will be evaluated through the Single-Leg Balance Test, Single-Leg Forward Hop Test, and Weight-Bearing Lunge Test. In addition, pain will be assessed using the VAS (Visual Analog Scale), and functional status will be measured with the VISA-A questionnaire. By conducting a comparative analysis, this study aims to evaluate the effects of architecture-based loading relative to classical protocols, thereby offering a novel perspective for treatment.

In light of this information, the present randomized controlled experimental trial has been designed to compare the effects of a muscle architecture-based exercise program with the classical Alfredson protocol on muscle-tendon architecture, muscle strength and endurance, functional performance, and symptomatic outcomes in individuals diagnosed with non-insertional Achilles tendinopathy.

ELIGIBILITY:
Inclusion Criteria:

* Presence of pain and tenderness in the mid-portion of the Achilles tendon (2-6 cm proximal to the insertion) persisting for at least 3 months
* Clinical diagnosis of non-insertional Achilles tendinopathy
* Pain aggravated by physical activity
* Palpable tenderness localized to the mid-portion of the tendon
* Voluntary participation in the study with signed informed consent

Exclusion Criteria:

* Diagnosis of insertional Achilles tendinopathy
* History of surgery or fracture in the affected lower limb within the past 12 months
* Corticosteroid injection to the Achilles tendon within the past month
* Presence of systemic diseases (e.g., diabetes mellitus, rheumatoid arthritis)
* Presence of neurological disorders (e.g., peripheral neuropathy, central nervous system disorders)
* Prior experience with eccentric exercise protocols targeting the Achilles tendon
* Acute onset of symptoms suggestive of a tendon rupture

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2025-10-15 (Estimated); Primary Completion 2026-12-15 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength and Endurance - Cybex HUMAC/NORM Isokinetic Dynamometer | From enrollment to the end of treatment at 12 weeks
  Lower limb plantar flexor strength and endurance will be assessed using the Cybex HUMAC/NORM 2002 isokinetic dynamometer. Participants will be seated securely in the test chair, with trunk and pelvis stabilized by straps.The ankle joint will be aligned with the dynamometer axis at the lateral malleolus, starting in 0° plantargrade neutral. Range of motion will be set between 20° dorsiflexion and 30° plantar flexion, and participants will wear flat-soled shoes.
  Three test protocols will be applied:
  Soleus-dominant assessment: knee flexed at 80-90°, concentric mode, angular velocity 90°/s, 20 consecutive repetitions; outcome: peak torque (Nm) Eccentric-concentric assessment: knee extended, eccentric-concentric mode, velocity 90°/s, 3 maximal repetitions; outcome: peak torque (Nm).
  Combined gastrocnemius-soleus assessment: knee extended, concentric-concentric mode, velocity 180°/s outcome: peak torque (Nm).
Muscle and Tendon Architecture Measurements | From enrollment to the end of treatment at 12 weeks
  Muscle architecture of the medial and lateral gastrocnemius and soleus will be assessed with B-mode ultrasonography. Outcomes include fascicle length (cm), pennation angle (°), thickness (mm), cross-sectional area (cm²), and volume (cm³). Participants will be prone with standardized alignment; images will be acquired using a 5-12 MHz probe in longitudinal and transverse planes. Muscle thickness will be measured between aponeuroses, fascicle length measured directly or calculated, pennation angle determined from fascicle-aponeurosis intersection, CSA traced from transverse images, and volume calculated from serial CSA values. Image analysis will be performed using ImageJ. Achilles tendon will be evaluated with a 10-15 MHz probe in prone with slight knee flexion. Outcomes include tendon thickness (mm, 3 cm proximal to insertion), fibrillar organization scored qualitatively, and neovascularization graded via Power Doppler. All measurements will be obtained by blinded experienced examiner
Function - Victorian Institute of Sport Assessment-Achilles (VISA-A) | From enrollment to the end of treatment at 12 weeks
  The VISA-A is an 8-item, self-reported questionnaire specifically developed to assess symptoms related to Achilles tendinopathy. Scores range from 0 to 100, with higher values indicating better clinical status. The scale has been demonstrated to be a valid and reliable tool for evaluating the clinical severity of Achilles tendinopathy. The Turkish version (VISA-A-Tr) has also shown high test-retest reliability and acceptable internal consistency, confirming its suitability for use in this population.
Muscle Elasticity - Myoton PRO | From enrollment to the end of treatment at 12 weeks
  Muscle and tendon elasticity will be assessed with the MyotonPRO device in prone position with ankles in neutral. The probe applies a brief mechanical impulse, and five measurements per site will be averaged. Measurements will be obtained at the medial gastrocnemius, lateral gastrocnemius, soleus, and Achilles tendon. Separate outcomes will be reported for each parameter: frequency (Hz), stiffness (N/m), decrement (logarithmic), creep (µm/N), and relaxation time (ms). This method provides reliable and reproducible data on tissue mechanical properties.
Single Leg Forward Hop Distance (cm) | From enrollment to the end of treatment at 12 weeks
  Participants will stand on the test leg and perform a maximal forward hop, landing on the same leg with controlled balance. One practice trial will be allowed, followed by three valid attempts, with the longest distance in centimeters (cm) used for analysis. To be considered valid, participants must maintain balance for at least two seconds after landing. Contact with the opposite leg, instability, or multiple hops will invalidate the trial. Arm movement is permitted. Rest intervals will include 30 seconds between attempts and 2 minutes between tests. This test is applied to evaluate lower limb functional performance and inter-limb symmetry. Previous studies have demonstrated excellent reliability and low measurement error for this assessment.
Single Leg Stance Balance Time (seconds) | From enrollment to the end of treatment at 12 weeks
  Participants will attempt to maintain balance barefoot on one leg while standing on a firm surface. The outcome is recorded as balance duration in seconds (s). Movement of the test leg or ground contact by the contralateral leg invalidates the trial. Testing is performed under both eyes-open and eyes-closed conditions. Each leg is tested three times with up to 60 seconds per trial and 1-minute rest intervals. The best performance under each condition is used for analysis. This measure reflects static balance ability.
Ankle Mobility - Weight-Bearing Lunge Test | From enrollment to the end of treatment at 12 weeks
  Ankle dorsiflexion range of motion will be assessed using the weight-bearing lunge test. Participants will stand barefoot facing a wall in a lunge position with the test limb in front. Without lifting the heel, they will move the knee forward until it touches the wall, and the maximum distance from the wall to the tip of the great toe will be measured in centimeters with a tape measure. Each limb will be tested three times, and the best value will be recorded for analysis. A 30-second rest will be provided between trials. Standardized verbal instructions will be given, and pain will be monitored using the Numeric Rating Scale. This method is considered a valid and reliable measure of ankle dorsiflexion mobility.

SECONDARY OUTCOMES:
Pain - Numeric Rating Scale (NRS) | From enrollment to the end of treatment at 12 weeks
  Pain intensity will be assessed using the 3-stage Numeric Rating Scale. Participants will rate their "worst pain," "least pain," and "current pain" experienced in the past 24 hours on a scale from 0 to 10. The mean of these three values will be recorded as the overall pain score. The NRS is a widely used, valid, and reliable tool for quantifying pain in musculoskeletal conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul University, Istanbul, Fatih, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Al-Uzri, M., O'Neill, S., Watson, P., & Kelly, C. (2016). Reliability of isokinetic dynamometry of the plantarflexors in knee flexion and extension. Physiotherapy practice and research, 38(1), 49-57.
- [Background] O'Neill S, Barry S, Watson P. Plantarflexor strength and endurance deficits associated with mid-portion Achilles tendinopathy: The role of soleus. Phys Ther Sport. 2019 May;37:69-76. doi: 10.1016/j.ptsp.2019.03.002. Epub 2019 Mar 9. PMID 30884279
- [Background] Del Bano-Aledo ME, Martinez-Paya JJ, Rios-Diaz J, Mejias-Suarez S, Serrano-Carmona S, de Groot-Ferrando A. Ultrasound measures of tendon thickness: Intra-rater, Inter-rater and Inter-machine reliability. Muscles Ligaments Tendons J. 2017 May 10;7(1):192-199. doi: 10.11138/mltj/2017.7.1.192. eCollection 2017 Jan-Mar. PMID 28717629
- [Background] Lauber B, Lichtwark GA, Cresswell AG. Reciprocal activation of gastrocnemius and soleus motor units is associated with fascicle length change during knee flexion. Physiol Rep. 2014 Jun 11;2(6):e12044. doi: 10.14814/phy2.12044. Print 2014 Jun 1. PMID 24920126
- [Background] Kwah LK, Pinto RZ, Diong J, Herbert RD. Reliability and validity of ultrasound measurements of muscle fascicle length and pennation in humans: a systematic review. J Appl Physiol (1985). 2013 Mar 15;114(6):761-9. doi: 10.1152/japplphysiol.01430.2011. Epub 2013 Jan 10. PMID 23305989
- [Background] Phillips B, Buchholtz K, Burgess TL. Gastrocnemius muscle architecture in distance runners with and without Achilles tendinopathy. S Afr J Sports Med. 2022 Jan 1;34(1):v34i1a12576. doi: 10.17159/2078-516X/2022/v34i1a12576. eCollection 2022. PMID 36815930
- [Background] Beyer R, Kongsgaard M, Hougs Kjaer B, Ohlenschlaeger T, Kjaer M, Magnusson SP. Heavy Slow Resistance Versus Eccentric Training as Treatment for Achilles Tendinopathy: A Randomized Controlled Trial. Am J Sports Med. 2015 Jul;43(7):1704-11. doi: 10.1177/0363546515584760. Epub 2015 May 27. PMID 26018970
- [Background] Alfredson H, Pietila T, Jonsson P, Lorentzon R. Heavy-load eccentric calf muscle training for the treatment of chronic Achilles tendinosis. Am J Sports Med. 1998 May-Jun;26(3):360-6. doi: 10.1177/03635465980260030301. PMID 9617396